CLINICAL TRIAL: NCT03605914
Title: Are NSAIDs Effective Enough for Postoperative Pain Control After Functional Endoscopic Sinus Surgery and Septoplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Martin J Citardi, MD, Professor and Chairman, Department of Otorhinolaryngology - Head and Neck Surgery, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-18-0242
Record Dates: First submitted 2018-07-04; First posted 2018-07-30 (Actual); Results first posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Pain Control After Functional Endoscopic Sinus Surgery and Septoplasty
MeSH Terms: interventions — Diclofenac; oxycodone-acetaminophen

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- NSAID (Experimental): The non-steroidal anti-inflammatory drug (NSAID) used in this study is diclofenac.
  Interventions: Drug: diclofenac
- opioid (Active Comparator): The Opioid used in this study is Norco. Norco is a combination medication that contains both an opioid pain reliever (hydrocodone) and a non-opioid pain reliever (acetaminophen).
  Interventions: Drug: Norco

INTERVENTIONS:
Drug: diclofenac — The non-steroidal anti-inflammatory drug (NSAID) used in this study is diclofenac.
  Arms: NSAID
Drug: Norco — The opioid used in this study is Norco. Norco is a combination medication that contains both an opioid pain reliever (hydrocodone) and a non-opioid pain reliever (acetaminophen).
  Other Names: Hydrocodone-Acetaminophen combination medication
  Arms: opioid

SUMMARY:
The purpose of this study is to compare the level of pain control in patients receiving non-steroidal anti-inflammatory drugs (NSAIDs) to those receiving opioids in the postoperative period after endoscopic sinus surgery (ESS) and/or septoplasty.

ELIGIBILITY:
Inclusion Criteria:

* english speaking
* candidates for endoscopic sinus surgery as determined by medical necessity by the treating rhinologist
* scheduled for surgery at Texas Sinus Institute

Exclusion Criteria:

* allergy to either NSAIDs or opioids
* contraindication to NSAIDs (ex. gastritis, chronic kidney disease)
* surgical plan exceeding basic endoscopic sinus surgery
* use of anticoagulation
* the presence of any pain disorder
* the current usage of any analgesic medication
* history of opioid addiction
* pregnancy
* history of chronic pain or fibromyalgia
* current daily use of NSAIDs, acetaminophen, opioids or other analgesics (pregabalin, tramadol, etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Citardi, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NSAID | Opioid
Started | 57 | 43
Completed Day 1 Assessment | 31 | 26
Completed Day 2 Assessment | 32 | 27
Completed Day 3 Assessment | 31 | 28
Completed Day 5 Assessment | 30 | 24
Completed | 30 | 24
Not Completed | 27 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NSAID | Opioid | Total
Number analyzed (Participants) | 57 | 43 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (15.7) | 46.2 (15.3) | 45.7 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 17 | 37
  Male | 37 | 26 | 63
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 57 | 43 | 100
Number of participants with history of anxiety [Count of Participants; unit: Participants] | 6 | 3 | 9
Number of participants with history of depression [Count of Participants; unit: Participants] | 4 | 3 | 7
Number of participants with history of migraine [Count of Participants; unit: Participants] | 5 | 3 | 8
Number of participants with history of temporomandibular joint (TMJ) dysfunction [Count of Participants; unit: Participants] | 0 | 0 | 0
Number of participants with history of fibromyalgia [Count of Participants; unit: Participants] | 0 | 0 | 0
Number of participants with history of pain disorder [Count of Participants; unit: Participants] | 0 | 0 | 0
Number of participants currently on pain medication [Count of Participants; unit: Participants] | 1 | 0 | 1
Number of participants currently on opioid [Count of Participants; unit: Participants] | 0 | 0 | 0
Number of participants currently on NSAID [Count of Participants; unit: Participants] | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Pain Score as Assessed by a 100mm Visual Analogue Scale (VAS)
Description: The range of scores on the VAS is 0 to 100, with 100 being the highest level of pain.
Time Frame: 24 hours (day 1 after operation)
Population: Data was not collected for 26 in the NSAID arm and 17 in the opioid arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NSAID | Opioid
Number analyzed (Participants) | 31 | 26
units on a scale | 30.2 (25.3) | 40.7 (29.2)

2. Secondary Outcome: Pain Score as Assessed by a 100mm Visual Analogue Scale (VAS)
Description: The range of scores on the VAS is 0 to 100, with 100 being the highest level of pain.
Time Frame: 48 hours (day 2 after operation)
Population: Data was not collected for 25 in the NSAID arm and 16 in the opioid arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NSAID | Opioid
Number analyzed (Participants) | 32 | 27
units on a scale | 24.2 (25.1) | 28.3 (23.4)

3. Secondary Outcome: Pain Score as Assessed by a 100mm Visual Analogue Scale (VAS)
Description: The range of scores on the VAS is 0 to 100, with 100 being the highest level of pain.
Time Frame: 72 hours (day 3 after operation)
Population: Data was not collected for 26 in the NSAID arm and 15 in the opioid arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NSAID | Opioid
Number analyzed (Participants) | 31 | 28
units on a scale | 22.9 (20.4) | 27.9 (21.9)

4. Secondary Outcome: Pain Score as Assessed by a 100mm Visual Analogue Scale (VAS)
Description: The range of scores on the VAS is 0 to 100, with 100 being the highest level of pain.
Time Frame: 120 hours (day 5 after operation)
Population: Data was not collected for 27 in the NSAID arm and 19 in the opioid arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NSAID | Opioid
Number analyzed (Participants) | 30 | 24
units on a scale | 17.2 (20.3) | 18.9 (18.8)

5. Secondary Outcome: Number of Participants With Bleeding Complications
Description: Bleeding complications are defined as complications necessitating a trip to the emergency room or requiring intervention for epistaxis.
Time Frame: 5 days after operation
Population: Data was not collected for 27 in the NSAID arm and 19 in the opioid arm.
Measure: Count of Participants; unit: Participants
Arm/Group | NSAID | Opioid
Number analyzed (Participants) | 30 | 24
Participants | 0 | 0

6. Secondary Outcome: Number of Participants With Constipation
Time Frame: 5 days after operation
Population: No data were collected for this outcome measure.
Arm/Group | NSAID | Opioid
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants With Nausea or Vomiting
Time Frame: 5 days after operation
Population: No data were collected for this outcome measure.
Arm/Group | NSAID | Opioid
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 5 days
Arm/Group | NSAID | Opioid
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/43
Other Adverse Events (participants affected / at risk) | 0/57 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-26): https://cdn.clinicaltrials.gov/large-docs/14/NCT03605914/Prot_SAP_000.pdf